CLINICAL TRIAL: NCT07011992
Title: A Phase 1, Open-label, 1-Sequence Crossover, Drug-drug Interaction Study to Assess the Effect of Repeated Doses of BPN14770 on the Pharmacokinetics of Rosuvastatin in Healthy Adult Participants
Brief Title: A Study to Assess the Effects of BPN14770 on Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2413A4111
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: BPN14770; Rosuvastatin; Pharmacokinetics
MeSH Terms: interventions — Rosuvastatin Calcium; BPN14770

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BPN14770 (Experimental): Participants will receive rosuvastatin and BPN14770.
  Interventions: Drug: Rosuvastatin; Drug: BPN14770

INTERVENTIONS:
Drug: Rosuvastatin — Oral tablet
Drug: BPN14770 — Oral capsule
  Other Names: Zatolmilast

SUMMARY:
The primary objective of this study is to investigate the effects of BPN14770 on the pharmacokinetics of the breast cancer resistance protein and organic anion transporting polypeptide 1B1 substrate rosuvastatin in healthy adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Overtly healthy as determined by medical evaluation including medical history, medical examination, laboratory tests, vital sign measurements, and 12-lead electrocardiogram at screening and on admission or participants whose laboratory values exceed the institutional reference range but deemed not clinically significant by the investigator in consideration of safety
* Body mass index ≥18.5 and <32.0 kilograms/meter squared
* All female participants must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations)

Key Exclusion Criteria:

* Presence or history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological, or ophthalmological (that is, increased intraocular pressure) disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data per the investigator's assessment
* Known history of allergic reaction to multiple medications and/or severe allergic reaction to any food or environmental allergens
* Prior use of rosuvastatin that was discontinued for tolerability or adverse events
* Received ≥4 types of investigational study interventions within 12 months prior to administration of study intervention
* Positive drug or alcohol screen test result at screening or upon admission
* Use of cannabis (medical or recreational), tobacco, or nicotine-containing products (including e-cigarettes, pipe tobacco, cigar, chewing tobacco, nicotine patch, and nicotine gum) within 6 months prior to admission

Note: Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-07-18 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Rosuvastatin | Days 1 and 11 (pre-dose, up to 72 hours post-dose)
Time to Maximum Plasma Concentration (Tmax) of Rosuvastatin | Days 1 and 11 (pre-dose, up to 72 hours post-dose)

SECONDARY OUTCOMES:
Cmax of BPN14770 | Day 11 (pre-dose, up to 72 hours post-dose)
Tmax of BPN14770 | Day 11 (pre-dose, up to 72 hours post-dose)
Cmax of Coproporphyrin I | Days 1 and 11 (pre-dose, up to 72 hours post-dose)
Tmax of Coproporphyrin I | Days 1 and 11 (pre-dose, up to 72 hours post-dose)
Number of Participants Experiencing Treatment-emergent Adverse Events | Day 1 through Day 21

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Clinical Research, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No